CLINICAL TRIAL: NCT03017391
Title: Feasibility Study to Compare 2 Strategies of Treatment Algorithm for Treating Nausea and or Vomiting in the Palliative Phase of Cancer Care
Brief Title: Treatment Algorithm for Nausea and Vomiting in the Palliative Phase
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVS01
Record Dates: First submitted 2016-04-21; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-12

CONDITIONS: Nausea; Vomiting; Cancer
Keywords: palliative care; palliative medicine; palliative
MeSH Terms: conditions — Nausea; Vomiting; Neoplasms | interventions — Metoclopramide; Granisetron; Dexamethasone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- algorithm 1 first metoclopramide (Active Comparator): metoclopramide 10 mg tablets 3x daily orally and in those patients that cannot swallow tablets the medication will be substituted by suppositories 10 mg 3x daily rectally. In case of failure, granisetron patch 3.1mg/24 hours will be added to the treatment and a loading dose of 2 mg granisetron oral if the patient can swallow. In case of toxicity metoclopramide will be stopped. In case of failure of the combination (second step) or toxicity, an oral dose of dexamethasone 8 mg will be added daily.
  Interventions: Drug: metoclopramide; Drug: granisetron; Drug: Dexamethasone; Drug: Granisetron 2Mg Tablet
- algorithm 2 first granisetron (Active Comparator): granisetron patch 3.1 mg/24 hours will be offered to the patient, and a loading dose of 2 mg granisetron oral if the patient can swallow In case of failure, metoclopramide 10 mg tablets 3x daily orally will be added and in those patients that cannot swallow tablets the oral medication will be substituted with rectal suppositories 10 mg. The granisetron patch will only be withdrawn from patients that suffer from clinically relevant toxicity. Metoclopramide will then be administered.
  In the case of secondary failure or toxicity, dexamethasone 8 mg orally daily will be added.
  Interventions: Drug: metoclopramide; Drug: granisetron; Drug: Dexamethasone; Drug: Granisetron 2Mg Tablet

INTERVENTIONS:
Drug: metoclopramide — metoclopramide 10 mg tablets 3x daily orally or suppositories 10 mg 3x daily rectally, use until toxicity
Drug: granisetron — granisetron patch 3.1mg/24 hours, use until toxicity
  Other Names: Sancuso
Drug: Dexamethasone — dexamethasone 8 mg, last step in both algorithms
Drug: Granisetron 2Mg Tablet — granisetron 2 mg loading dose

SUMMARY:
Nausea and vomiting are frequently occurring problems in the palliative phase of patients with cancer. Between 20-50% of them regularly suffer from nausea, retching or vomiting. Often the cause of nausea and vomiting is multifactorial and symptomatic treatment is necessary.

Potential drugs for symptomatic anti-nausea therapy are metoclopramide, serotonin antagonists, the combination of both and dexamethasone as rescue medication in case of failure. There is no data that depicts which strategy is the best. This study will be conducted to unravel which treatment algorithm is most successful.

DETAILED DESCRIPTION:
Nausea and vomiting are frequently occurring problems in the palliative phase of patients with cancer. Between 20-50% of them regularly suffer from nausea, retching or vomiting. Often the cause of nausea and vomiting is multifactorial and symptomatic treatment is necessary.

Potential drugs for symptomatic anti-nausea therapy are metoclopramide, serotonin antagonists, the combination of both and dexamethasone as rescue medication in case of failure. There is no data that depicts which strategy is the best. This study will be conducted to unravel which treatment algorithm is most successful: 1 to start with metoclopramide, to add a serotonin antagonist (granisetron transdermal patch and 2 milligram granisetron oral loading dose if the patient can swallow) in case of failure and to add dexamethasone as rescue medication versus 2 an algorithm to start with a serotonin antagonist (granisetron transdermal patch and 2 milligram granisetron oral loading dose if the patient can swallow), to add metoclopramide in case of failure and to add dexamethasone as rescue medication. Granisetron plaster is a new formulation of a well known serotonin antagonist and might be useful especially within the patient group in the palliative phase.

The questions are:

Is it feasible to compare treatment algorithms for symptomatic treatment of nausea and vomiting in palliative cancer patients? And is a stepwise symptomatic treatment algorithm to manage nausea and vomiting using metoclopramide or granisetron transdermal patch as a start medication effective in palliative patients in at least one of both treatment arms? Patients will be asked to complete the QLQC30 and ESAS on different moments during the study. Besides, they will be asked to complete a diary for nausea severity (NRS scale 0-10) and for the frequency of vomiting and retching twice daily.

Success of a treatment algorithm is defined as nausea is < 3 on NRS or a decrease of >2 on NRS for nausea combined with an absence of vomiting or retching in the last 3 days. Incomplete success is defined as nausea of 3 on NRS during one occasion of the last 3 days before the end of study but less than 4, no more than one retching a day during that period and absence of vomiting. Complete failure is defined as nausea of 4 or more on an NRS during the last 3 days or more than one retching daily or any vomiting or in case the patient has stopped all medication due to side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years or older in the palliative phase and
* who suffer from nausea or vomiting with a rating on a numeric rating scale (NRS) of more than 2 and
* have a wish to be treated and
* where no treatable cause is assignable

Exclusion Criteria:

* Patients not able to sign informed consent.
* Patients with known contra-indications for metoclopramide, 5HT-3 antagonists or dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
NRS nausea | 15 days
  response defined as NRS <3 or decrease of more than 2 on NRS and absence of vomiting or retching in the last 3 days

SECONDARY OUTCOMES:
days from T0 to control | two weeks
  The time from T0 until the moment that nausea and vomiting/retching is in control

OTHER OUTCOMES:
feasibility | 6 months
  number of included patients a 6 months period
comparison of starting metoclopramide to starting with granisetron | 6 months
  response defined as NRS <3 or decrease of more than 2 on NRS and absence of vomiting or retching in the last 3 days
quality of life | 15 days
  QLQC30 scale
adverse events | 14/15 days
  diary adverse events

CONTACTS AND LOCATIONS:
Overall Officials: C.A.H.H.V.M. Verhagen, M.D. Ph.D., Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No